CLINICAL TRIAL: NCT07397078
Title: Moni-Patch Temperature Monitoring Patch System Clinical Accuracy Validation
Brief Title: Clinical Accuracy Validation of the Moni-Patch Temperature Monitoring Patch System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murata Vios, Inc. (Industry)
Collaborators: Sonoma State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MPS2_01
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Body Temperature; Febrile
Keywords: Core body temperature
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Concurrent Monitoring (Experimental): Subjects wear Moni-Patch on the neck and tympanic sensor in the ear for concurrent continuous temperature monitoring for 15 minutes after stabilization.
  Interventions: Device: Moni-Patch Temperature Monitoring Patch System

INTERVENTIONS:
Device: Moni-Patch Temperature Monitoring Patch System — Wireless neck-applied Sensor paired with a Receiver via Bluetooth; heat flux and thermistor-based estimation of core temperature; sampling every 30 seconds.
  Other Names: MP-P20U (Sensor); MP-D20U (Receiver)

SUMMARY:
Moni-Patch Temperature Monitoring Patch System, a non-invasive, continuous temperature monitoring device designed to estimate core body temperature by applying a Sensor to the neck.

This clinical accuracy validation study aims to verify the accuracy and repeatability of the Moni-Patch compared with an FDA-cleared continuous tympanic temperature monitoring device used as the clinical reference.

Main objectives of this study are; To verify that the Moni-Patch and the reference device(tympanic) demonstrate acceptable agreement, as defined by Bland-Altman Analyses (bias within ±0.4°C and limits of agreement between -1.0°C and 1.0°C).

To verify the consistency and repeatability of temperature measurements obtained from the Moni-Patch during continuous monitoring.

DETAILED DESCRIPTION:
This study is conducted in accordance with ISO 80601-2-56:2017, which outlines definitions for temperature-measuring devices, age groups, required sample sizes, fever definitions, procedural flow, and statistical methods for clinical performance evaluation.

All subjects undergo temperature measurement using the reference device(Tympanic) and the investigational device (Moni-Patch Temperature Monitoring Patch System). The Moni-Patch Sensor is applied to the neck and paired with the Receiver, while the tympanic probe is positioned and sealed in the ear canal.

Each subject participates in a continuous 15-minute temperature monitoring session, during which both devices collect temperature values concurrently every 30 seconds.

Environmental temperature and humidity are also recorded during the session.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 7 years
* Agree to Sensor placement on the neck and ear

Exclusion Criteria:

* Ear conditions contraindicating tympanic probe; skin issues at placement sites
* Antipyretic use within 120 minutes; inability to position neck Sensor over carotid
* Inability to seal tympanic sensor; tympanic membrane not visually confirmed

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between Moni-Patch™ Core Temperature Monitoring Patch System and Continuous Tympanic Temperature (Ttym) Measurements | 15-minute continuous temperature monitoring period following a minimum 30-minute sensor acclimation period (per subject).
  Agreement will be quantified using the mean temperature difference (bias; °C) and Limits of Agreement (LOA; °C) between the Moni-Patch™ Temperature Monitoring Patch System and the comparative FDA-cleared continuous tympanic thermometer (Ttym).
  Paired temperature measurements (Moni-Patch vs. Ttym) collected every 30 seconds during continuous monitoring will be analyzed using Bland-Altman methodology.
  Name of Measurement: Core body temperature difference
  Measurement Tool(s):
  Moni-Patc Temperature Monitoring Patch System FDA-cleared continuous tympanic temperature monitoring device (Ttym)
  Unit of Measure: Degrees Celsius (°C) Analysis Method: Bland-Altman bias and 95% limits of agreement

CONTACTS AND LOCATIONS:
Locations (1):
- Murata Vios, Woodbury, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
De-identified instrument data will be analyzed by the Sponsor; no public IPD sharing is planned.